CLINICAL TRIAL: NCT07158528
Title: An RCT Comparing Coronally Advanced Flap (CAF) and Tunneled Coronally Advanced Flap (TCAF) in Combination With a Soft Tissue Graft for Multiple Recessions Coverage in the Maxilla.
Brief Title: Comparing CAF and TCAF With Soft Tissue Grafting for Treating Multiple Recessions in the Maxilla.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ONZ-2025-0158
Record Dates: First submitted 2025-08-28; First posted 2025-09-08 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Gingival Recession Generalized Moderate; Gingival Recession Localized Moderate; Gingival Recession, Generalized; Gingival Recession, Localized; Gingival Recession, Plastic Surgery; Gingival Recessions; Gingival Recession, Mucogingival Surgery
Keywords: TCAF; CAF; tunneled coronally advanced flap; coronally advanced flap; maxilla; multiple recessions; MAGR; multiple adjacent gingival recessions
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TCAF + CTG (Active Comparator): Tunneled coronally advanced flap with a connective tissue graft.
  Interventions: Procedure: tunneled coronally advanced flap with a connective tissue graft
- CAF + CTG (Active Comparator): Coronally advanced flap with a connective tissue graft.
  Interventions: Procedure: coronally advanced flap with connective tissue graft

INTERVENTIONS:
Procedure: coronally advanced flap with connective tissue graft — The gum at the recession site is elevated and repositioned higher, combined with a connective tissue graft.
  Other Names: CAF + CTG
  Arms: CAF + CTG
Procedure: tunneled coronally advanced flap with a connective tissue graft — The gum at the recession site is undermined, only partially detached, and repositioned higher, combined with a connective tissue graft.
  Other Names: TCAF + CTG
  Arms: TCAF + CTG

SUMMARY:
Multiple techniques can be used for recession coverage. The most common techniques are: tunnel technique (T), coronally advanced flap (CAF) or a combination of both (TCAF). Tunnel and coronally advanced flap are frequently used in clinical practice, whereas the combined technique is a relatively recently developed surgical approach.

This randomized controlled trial compares CAF and TCAF to determine which technique provides better root coverage for receding gums at multiple adjacent teeth in the upper jaw. The main question it aims to answer is:

- What is the average root coverage achieved with each technique in the short and long term? This may be clinically relevant because covering gum recession can reduce tooth sensitivity, improve aesthetics and make oral hygiene easier.

Researchers will compare the coronally advanced flap (CAF = the gum is detached and repositioned higher) with the tunneled coronally advanced flap (TCAF = the gum is undermined, only partially detached and repositioned higher). In both techniques, a small piece of tissue is removed from the palate, which is used to cover the recession. The purpose of the connective tissue graft under the flap/tunnel is to increase thickness and provide support.

Participants will:

* Undergo surgery (CAF or TCAF, randomly assigned) to cover recessions
* Attend regular check-ups for up to 10 years after surgery
* Keep a postoperative journal (recording medication use, pain levels, tooth sensitivity, etc.)

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Good oral hygiene
* Presence of multiple gingival recessions in the maxilla
* Good general health

Exclusion Criteria:

* Smoker
* Pregnant women (assessed at each visit; if the patient becomes pregnant during follow-up, radiographs will not be taken)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-08-18 (Actual); Primary Completion 2037-12-31 (Estimated); Study Completion 2037-12-31 (Estimated)

PRIMARY OUTCOMES:
mean root coverage | From enrollment up to ten years after surgical treatment.
  The average percentage of previously exposed tooth surface that becomes covered by gingival tissue following a root coverage procedure.

SECONDARY OUTCOMES:
complete root coverage | From enrollment up to ten years after surgical treatment.
  The percentage of teeth for which the previously exposed root surface is completely covered by gingival tissue following the surgical procedure. These teeth show no visible recession after healing.
pocket depth | From enrollment up to ten years after surgical treatment.
  The distance from the gingival margin to the bottom of the sulcus measured by use of a periodontal probe.
recession reduction | From enrollment up to ten years after surgical treatment.
  The change in the amount of exposed root surface after the root coverage procedure.
width of keratinized tissue | From enrollment up to ten years after surgical treatment.
  The distance from the mucogingival junction to the free gingival margin. It includes free and attached gingival tissue, measured by use of a periodontal probe.
gingival thickness | From enrollment up to ten years after surgical treatment.
  Thickness of the gingival tissue, measured 1-2 mm apical to the gingival margin.
phenotype | From enrollment up to ten years after surgical treatment.
  Gingival phenotype is classified as thin, thick or combined.
treatment time | Only measured during surgery in minutes.
  Time in minutes from the first incision up to the last suture.
post-operative pain at the donor site | From one week post-operative up to three months post-operative.
  Post-operative pain at the donor site will be assessed by the patient using the Visual Analogue Scale (VAS), ranging from 0 (no pain) to 10 (worst imaginable pain). A higher score indicates greater pain experienced by the patient.
post-operative pain at the recession site | From one week post-operative up to three months post-operative.
  Post-operative pain at the recession site will be assessed by use of the Visual Analogue Scale (VAS), ranging from 0 (no pain) to 10 (worst imaginable pain). A higher score indicates greater pain experienced by the patient.
number of analgesics | From one week post-operative up to two weeks post-operative.
  The number of pain medication tablets consumed by the patient to manage post-operative pain.
score of the aesthetic outcome | From six months post-operative up to ten years post-operative.
  Aesthetic satisfaction will be based on root coverage and color match. Aesthetic satisfaction at the recession site will be assessed by use of the Visual Analogue Scale (VAS), ranging from 0 (aesthetic satisfaction not achieved) to 10 (aesthetic satisfaction fully achieved). A higher score indicates greater satisfaction.
root sensitivity | From one week pre-operative up to ten years post-operative.
  Root sensitivity is assessed by use of the Visual Analogue Scale (VAS), ranging from 0 (no sensitivity) to 10 (extreme sensitivity), based on a tactile test with controlled air flow. A higher score indicates that the patient experiences greater sensitivity.
willingness to retreatment | From three months post-operative up to two years post-operative.
  A patient's willingness to undergo retreatment based on their previous experience with the procedure. It is assessed by the use of the Visual Analogue Scale ranging from 0 (not willing at all) to 10 (extremely willing). A patient reporting a higher score indicates greater willingness.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Periodontology and Implantology of Ghent University, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: No